CLINICAL TRIAL: NCT02416180
Title: An Open-label Study Investigating Critical and Overall Errors Following 14 Days of Treatment With SERETIDE Metered Dose Inhaler (EVOHALER) in Adult Subjects With Controlled Asthma Currently Using the SERETIDE DISKUS Inhaler
Brief Title: Study to Evaluate Handling Errors in Usage of SERETIDE® Metered Dose Inhaler (MDI) (EVOHALER®) by Adult Subjects Currently Using the SERETIDE DISKUS® Inhaler
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201909
Record Dates: First submitted 2015-04-09; First posted 2015-04-14 (Estimated); Results first posted 2016-07-07 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Asthma
Keywords: EVOHALER; Asthma; SERETIDE; DISKUS Inhaler; MDI
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SERETIDE EVOHALER (Experimental): Subjects will switch from their current usual maintenance treatment of SERETIDE via DISKUS Inhaler to an equivalent dose of SERETIDE via the MDI (EVOHALER) at Visit 1. Subjects will use the MDI as 2 inhalations twice daily for approximately 14 days. Subjects will revert back to using SERETIDE DISKUS Inhaler again from Visit 2 (after 14 days) starting with the next scheduled dose.
  Interventions: Device: SERETIDE MDI; Device: Placebo DISKUS Inhaler; Device: Placebo MDI

INTERVENTIONS:
Device: SERETIDE MDI — Commercially available SERETIDE MDI (EVOHALER) containing fluticasone propionate/salmeterol. Subjects will use MDI as 2 inhalations twice daily at the dose equivalent to their usual maintenance treatment of SERETIDE via DISKUS Inhaler.
Device: Placebo DISKUS Inhaler — Placebo dry powder inhaler to be used to demonstrate the use of DISKUS inhaler at Visit 1
Device: Placebo MDI — Clear liquid propellant inhaler to be used to demonstrate the use of MDI at Visit 2

SUMMARY:
This study aims to explore the potential impact of switching inhalers by assessing the handling error rate (critical and non-critical) in controlled asthmatics currently treated with, and using correctly, SERETIDE via the DISKUS Inhaler who are switched to receiving SERETIDE via the Metered Dose Inhaler (MDI) (EVOHALER) without training by a Healthcare Professional (HCP).

This will be a descriptive, multi-centre, open-label, non randomized 14 day study assessing MDI technique in subjects with controlled asthma (Asthma Control Test [ACT] score >= 20 at Visit 1) currently treated with, and able to use correctly, SERETIDE via the DISKUS Inhaler. All the eligible subjects will be switched to an equivalent dose of SERETIDE via the MDI. Subjects will need to use the MDI inhaler in accordance the accompanying patient information leaflet (to be read prior to use) for approximately 14 days. No instruction, coaching or comment on inhaler technique will be provided by the HCP. MDI technique of subjects will be assessed at Visit 2 (after 14 days) and the errors will be recorded. Subject will revert back to using their SERETIDE DISKUS inhaler again from Visit 2. Subjects will be followed up by telephone for approximately 1 week after Visit 2.

A maximum of 110 subjects will be enrolled such that approximately 100 evaluable subjects complete the study. The total duration of the study for each subject will be approximately 21 days.

SERETIDE, EVOHALER and DISKUS are registered trademarks of the GlaxoSmithKline (GSK) group of companies

ELIGIBILITY:
Inclusion Criteria:

* >=18 years of age at the time of informed consent.
* A diagnosis of asthma as defined by the National Institutes of Health, 2007.
* Must be currently treated with SERETIDE via the DISKUS Inhaler and have been maintained on this dose for 3 months prior to Visit 1.
* Have controlled asthma defined as a total ACT score >= 20
* Must be able to use their DISKUS inhaler correctly. Correct use is defined as making no critical errors during the assessment of DISKUS inhaler use at Visit 1.
* Male
* Female subject is eligible to participate if she is not pregnant (as confirmed by a negative urine human chorionic gonadotrophin [hCG] test), not lactating, and at least one of the following conditions applies: 1. Non-reproductive potential defined as: Pre-menopausal females with one of the following; documented tubal ligation, documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, hysterectomy, documented bilateral Oophorectomy. Postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone [FSH] and estradiol levels consistent with menopause). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment. 2. Reproductive potential and agrees to follow one of the options listed below in the GSK modified list of highly effective methods for avoiding pregnancy in females of reproductive potential (FRP) requirements from 30 days prior to the first dose of study medication and until after the last dose of study medication and completion of the follow-up contact.

GSK modified list of highly effective methods for avoiding pregnancy in FRP: a. Contraceptive subdermal implant that meets the standard operating procedure (SOP) effectiveness criteria including a <1percent rate of failure per year, as stated in the product label. b. Intrauterine device or intrauterine system that meets the SOP effectiveness criteria including a <1 percent rate of failure per year, as stated in the product label. c. Oral Contraceptive, either combined or progestogen alone. d. Injectable progestogen. e. Contraceptive vaginal ring. f. Percutaneous contraceptive patches. g. Male partner sterilization with documentation of azoospermia prior to the female subject's entry into the study, and this male is the sole partner for that subject. h. Male condom combined with a vaginal spermicide (foam, gel, film, cream, or suppository). GSK modified list of highly effective methods for avoiding pregnancy in FRP does not apply to FRP with same sex partners, when this is their preferred and usual lifestyle or for subjects who are and will continue to be abstinent from penile-vaginal intercourse on a long term and persistent basis. These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and protocol.

Exclusion Criteria:

* Have a current diagnosis of chronic obstructive pulmonary disease (COPD)
* Have experienced an asthma exacerbation within 3 months of Visit 1 or a lower respiratory tract infection within 6 weeks of Visit 1. An exacerbation is defined as worsening asthma requiring any treatment other than rescue salbutamol. This includes requiring the use of systemic or inhaled corticosteroids and /or emergency room visit or hospitalisation.
* Other Concurrent Diseases: A subject must not have any clinically significant, uncontrolled condition or disease state (such as severe cardiovascular disorders or heart rhythm abnormalities, diabetes mellitus, thyrotoxicosis, uncorrected hypokalaemia or predisposition to low levels of serum potassium) that, in the opinion of the investigator (in consultation with the GSK Medical Monitor if required), would put the safety of the subject at risk through study participation or would confound the interpretation of the results if the condition/disease exacerbated during the study. Please refer to the SERETIDE Product Label for a full list of conditions for special warnings and precautions for use.
* Currently taking potent Cytochrome P450 3A4 (CYP 3A4) inhibitors
* Currently taking beta-blockers (selective and non-selective).
* Allergic to salmeterol, fluticasone propionate or to norflurane (HFA 134a) or to any other excipients.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than 4 investigational medicinal products within 12 months prior to the first dosing day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2015-06-18 (Actual); Primary Completion 2015-08-20 (Actual); Study Completion 2015-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- Germany (4):
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Neu-Isenburg, Hesse
  - GSK Investigational Site, Reinfeld, Schleswig-Holstein
  - GSK Investigational Site, Berlin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 201909 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 201909 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 201909 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 201909 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 201909 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 201909 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants with controlled asthma who were treated with fluticasone propionate/salmeterol via DISKUS inhaler, were asked to demonstrate how they currently use their DISKUS inhaler using a demonstration inhaler. Only participants who did not make any critical errors while demonstrating the inhaler technique were considered eligible for the study.
Groups:
- Fluticasone Propionate/Salmeterol MDI: Participants received fluticasone propionate/salmeterol via metered dose inhaler (MDI) for 14 days at a dose equivalent to their pre-study fluticasone propionate/salmeterol dose which was administered via DISKUS inhaler. Participants were instructed to read the fluticasone propionate/salmeterol MDI Patient Information Leaflet (PIL) and then to use the provided MDI in accordance with the PIL for approximately 14 days, in replacement of their DISKUS inhaler.
Period: Overall Study
Arm/Group | Fluticasone Propionate/Salmeterol MDI
Started | 111
Completed | 110
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Fluticasone Propionate/Salmeterol MDI: Participants received fluticasone propionate/salmeterol via MDI for 14 days at a dose equivalent to their pre-study fluticasone propionate/salmeterol dose which was administered via DISKUS inhaler. Participants were instructed to read the fluticasone propionate/salmeterol MDI PIL and then to use the provided MDI in accordance with the PIL for approximately 14 days, in replacement of their DISKUS inhaler.
Arm/Group | Fluticasone Propionate/Salmeterol MDI
Number analyzed (Participants) | 111
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.6 (16.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 47
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - Central/South Asian Heritage | 1
  Asian - Japanese Heritage | 1
  Asian - South East Asian Heritage | 2
  White - White/Caucasian/European Heritage | 106
  White - Mixed Race | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Making at Least One Critical Error After the First Assessment of Metered Dose Inhaler (MDI) Technique on Day 14
Description: Participant's inhaler use was assessed on Day 14 by the health care professional (HCP) against a predefined list of critical errors (CEs). Critical errors were defined as errors that were most likely to result in no or only minimal medication being inhaled. The participants were asked to demonstrate their usage of the MDI using a placebo demonstration MDI by HCP, critical or non-critical errors (N-CEs) and even no errors made by the participants while using the MDI were recorded. Critical errors in using the MDI were defined as: failure to remove the cap; failure to shake the device; failure to place the device in mouth; no dose actuated during an inhalation manoeuvre; dose coordination that was so poor that the patient was likely to have received no dose or only received minimal dose. 95% confidence interval (CI) is for the % of participants making at least one critical error after the first assessment of the MDI technique, and was calculated using the exact binomial distribution.
Time Frame: Day 14
Population: Intent to Treat (ITT) population: comprised of all participants who were screened and received at least one dose of study medication.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Fluticasone Propionate/Salmeterol MDI
Number analyzed (Participants) | 111
Percentage of Participants | 14 [8 to 21]

2. Secondary Outcome: Percentage of Participants Making at Least One Overall Error After the First Assessment of MDI Technique on Day 14.
Description: Inhaler use was assessed on Day 14 for overall errors. Overall errors included CEs or N-CEs. Demonstration of usage was with MDI and placebo, CE or N-CEs and even no errors were recorded. CEs were defined as: failure to remove the cap; failure to shake the device; failure to place the device in mouth; no dose actuated during an inhalation manoeuvre; dose coordination that was so poor that the patient was likely to have received no dose or only received minimal dose. N-CEs were defined as: failure to inhale within 5 seconds of shaking the device; no exhalation before an inhalation; the inhalation manoeuvre was not slow and/or was not deep; dose coordination was sub-optimal but patient likely to have received some dose; more than one actuation during an inhalation manoeuvre; did not hold breath. The exact 95% confidence interval is for percent of participants making at least one CE after the first assessment of the MDI technique, and was calculated using exact binomial distribution.
Time Frame: Day 14
Population: ITT population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Fluticasone Propionate/Salmeterol MDI
Number analyzed (Participants) | 111
Percentage of participants | 41 [31 to 50]

3. Secondary Outcome: Number of Health Care Professional (HCP) Instructions Required on Day 14
Description: Participant's inhaler use was assessed on Day 14 by the HCP against a predefined list of critical errors. If a participant made a critical error during this initial assessment, the HCP demonstrated the correct use of the inhaler to the participant and gave verbal instructions. The participant was then asked to demonstrate inhaler use. Any errors were recorded by the HCP. If the participant made a critical error then the HCP repeated the demonstration of inhaler use to the participant for a second time. If the participant continued to make a critical error in the use of the inhaler, the HCP demonstrated the correct use of the inhaler and gave verbal instructions one more time and the participant was then asked to demonstrate inhaler use. Instructions are only given to subjects who make a critical error. Any errors made after this final demonstration were recorded.
Time Frame: Day 14
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Fluticasone Propionate/Salmeterol MDI
Number analyzed (Participants) | 111
Participants
  0 Instruction | 96
  1 Instruction | 12
  2 Instructions | 2
  3 Instructions | 1

4. Secondary Outcome: Time Taken to Correctly Completing Inhaler Use at Day 14
Description: If a participant made a critical error during the initial assessment, the HCP demonstrated the correct use of the inhaler to the participant and gave verbal instructions. The HCP could have demonstrated the use of the inhaler a maximum of three times. Any errors made after this final demonstration were recorded. The time taken for the HCP to train the participant in the correct technique was recorded as T1: the time from when the participants started their demonstration of MDI use until they had completed their demonstration of MDI use (i.e., with no HCP support), T2: the time from when the HCP started to demonstrate/instruct device use until correct use was demonstrated by the participant (up to a maximum of three attempts only). T3 is defined as T1+T2, which is the time from when the participant started to demonstrate MDI use until correct use was demonstrated by the subject (up to a maximum of three attempts following demonstration by HCP).
Time Frame: Day 14
Population: ITT Population
Measure: Median (Full Range); unit: Minutes
Arm/Group | Fluticasone Propionate/Salmeterol MDI
Number analyzed (Participants) | 111
Minutes
  T1, n=96 | 1.14 [0.4 to 3.9]
  T2, n=15 | 3.23 [1.1 to 6.2]
  T3, n=111 | 1.25 [0.4 to 8.7]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious adverse events (SAE) were collected from the start of the study treatment until the follow-up contact (up to 23 days).
Description: AEs and SAEs were collected in the members of ITT Population, comprised of all participants in the treatment arm who gave informed consent and received at least one dose of study medication.
Arm/Group | Fluticasone Propionate/Salmeterol MDI
Serious Adverse Events (participants affected / at risk) | 1/111
Other Adverse Events (participants affected / at risk) | 4/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluticasone Propionate/Salmeterol MDI (N=111)
Perirectal abscess (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluticasone Propionate/Salmeterol MDI (N=111)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Asthenia (General disorders) | 1
Fatigue (General disorders) | 1
Hand-foot-and-mouth disease (Infections and infestations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.